CLINICAL TRIAL: NCT03026816
Title: Epidural Stimulation for Spinal Cord Injury
Brief Title: Epidural Stimulation After Neurologic Damage
Acronym: E-STAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Office of Higher Education (Other Government); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Hennepin Healthcare Research Institute (Other); Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUROSURG-2017-25478
Record Dates: First submitted 2017-01-01; First posted 2017-01-20 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Paraplegia, Complete
Keywords: epidural stimulation; spinal cord stimulation; autonomic dysfunction
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: All subjects will receive study intervention. Outcome assessments will be tested while the stimulator unit is on (intervention) and off (sham) during the study.
Masking Description: Masking is done during formal testing of BMCA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Epidural Spinal Cord Stimulation (Experimental): Epidural Spinal Cord Stimulation
  Interventions: Device: Epidural Spinal Cord Stimulation

INTERVENTIONS:
Device: Epidural Spinal Cord Stimulation — epidural spinal cord stimulator

SUMMARY:
This study will evaluate a method to optimize parameter settings in epidural spinal cord stimulation used to recover lower extremity volitional movement. The study will also characterize improvement in autonomic function (such as blood pressure control) and other functions related to spinal cord injury.

DETAILED DESCRIPTION:
Epidural spinal cord stimulation for the purpose of facilitating volitional movement is a new and novel neuromodulatory treatment. Epidural SCS has a long history of use for chronic pain with established medical device platforms. The purpose of this study is to investigate and establish the use of SCS for volitional movement. Specifically, establishing the disinhibitory effect of SCS in a greater population with inherent greater variability.

In addition to establishing the disinhibitory effect of SCS for cSCI, our study attempts to explore the parameter space of the spinal cord stimulator platforms in order to optimize stimulation settings for patients through the creation of a clinical decision support system (CDSS). Preliminary evidence suggests benefit to autonomic function, and this study also begins to explore the effects of SCS on cardiovascular function, urinary function, psychiatric outcomes, and quality of life, which all offer significant potential for patients suffering from chronic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Able to undergo the informed consent/assent process
* Stable, motor-complete paraplegia
* Discrete spinal cord injury between C6 and T10
* ASIA A or B Spinal Cord Injury Classification
* Medically stable in the judgement of the principal investigator
* Intact segmental reflexes below the lesion of injury
* Greater than 1 year since initial injury and at least 6 months from any required spinal instrumentation
* Willing to attend all scheduled appointments

Exclusion Criteria:

* Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery (e.g. cardiopulmonary issues)
* Inability to withhold antiplatelet/anticoagulation agents perioperatively
* Significant dysautonomia that would prohibit rehabilitation or assisted standing or any history of CVA or MI associated with autonomic dysreflexia. A single tilt table test with syncope, presyncope, or SBP < 50 or >200.
* Other conditions that would make the subject unable to participate in testing/rehabilitation in the judgement of the principal investigator
* Current and anticipated need for opioid pain medications or pain that would prevent full participation in the rehabilitation program in the judgement of the principal investigator
* Clinically significant mental illness in the judgement of the principal investigator
* Botulinum toxin injections in the previous 6 months
* Volitional movements present during EMG testing in bilateral lower extremities
* Unhealed spinal fracture
* Presence of significant contracture
* Presence of pressure ulcers
* Recurrent urinary tract infection refractory to antibiotics
* Current Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Volitional Response Index Magnitude | Months: 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15
  Brain Motor Control Assessment Volitional Response Index Magnitude

SECONDARY OUTCOMES:
Spinal cord stimulation for cardiovascular function | Over 12 months
  Systolic blood pressure measured during epidural stimulation (continuous)
Cerebrovascular Assessment Change | Months: 3, 6, 9
  Cerebral blood flow (CBF) during tilt table
Change in Visual Neurocognitive Assessment | Months: 3, 6, 9
  Stroop Test
Spinal cord stimulation optimization | Over 12 months
  Probit preference response surface obtained by serial force binary choice

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Shackleton C, Samejima S, Miller T, Sachdeva R, Parr A, Samadani U, Netoff T, Hocaloski S, Elliott S, Walter M, Darrow D, Krassioukov A. Effect of epidural spinal cord stimulation on female sexual function after spinal cord injury. Front Neurosci. 2023 Apr 5;17:1155796. doi: 10.3389/fnins.2023.1155796. eCollection 2023. PMID 37179555
- [Derived] Hoover C, Schuerger W, Balser D, McCracken P, Murray TA, Morse L, Parr A, Samadani U, Netoff TI, Darrow DP. Neuromodulation Through Spinal Cord Stimulation Restores Ability to Voluntarily Cycle After Motor Complete Paraplegia. J Neurotrauma. 2024 May;41(9-10):1163-1171. doi: 10.1089/neu.2022.0322. Epub 2023 Mar 22. PMID 36719784
- [Derived] Hoglund BK, Zurn CA, Madden LR, Hoover C, Slopsema JP, Balser D, Parr A, Samadani U, Johnson MD, Netoff TI, Darrow DP. Mapping Spinal Cord Stimulation-Evoked Muscle Responses in Patients With Chronic Spinal Cord Injury. Neuromodulation. 2023 Oct;26(7):1371-1380. doi: 10.1016/j.neurom.2022.10.058. Epub 2022 Dec 12. PMID 36517395
- [Derived] Darrow DP, Balser DY, Freeman D, Pelrine E, Krassioukov A, Phillips A, Netoff T, Parr A, Samadani U. Effect of epidural spinal cord stimulation after chronic spinal cord injury on volitional movement and cardiovascular function: study protocol for the phase II open label controlled E-STAND trial. BMJ Open. 2022 Jul 18;12(7):e059126. doi: 10.1136/bmjopen-2021-059126. PMID 35851008
- [Derived] Pena Pino I, Hoover C, Venkatesh S, Ahmadi A, Sturtevant D, Patrick N, Freeman D, Parr A, Samadani U, Balser D, Krassioukov A, Phillips A, Netoff TI, Darrow D. Long-Term Spinal Cord Stimulation After Chronic Complete Spinal Cord Injury Enables Volitional Movement in the Absence of Stimulation. Front Syst Neurosci. 2020 Jun 30;14:35. doi: 10.3389/fnsys.2020.00035. eCollection 2020. PMID 32714156
- See also: Clinical Trial Website — http://www.estand.org